CLINICAL TRIAL: NCT04164836
Title: The Effect of Suitable Nose Selection Using Rhinoscope on the Incidence and Severity of Epistaxis After Nasotracheal Intubation.
Brief Title: Effect of Nose Selection Using Rhnoscope on Epistaxis of Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AJIRB-MED-OBS-19-201
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Nasotracheal Intubation
Keywords: epistaxis; rhinoscope
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): nose selection will be done by random table
- rhinoscope group (Experimental): nose selection will be done by rhinoscopy
  Interventions: Diagnostic Test: rhinoscope

INTERVENTIONS:
Diagnostic Test: rhinoscope — more suitable nose for nasotracheal intubation will be selected based on the view of rhinoscope.
  Arms: rhinoscope group

SUMMARY:
Rhinoscope is useful to exam intranasal structure. This information could be utilized to select more suitable nose for nasotracheal intubation. Nastoracheal intubation using more patent nose could be associated with decrease of the development of epistaxis which is most common complication in nasotracheal intubation.

DETAILED DESCRIPTION:
Anterior rhinoscopy using rhinoscope is a simple way to view the intranasal structure, which allows you to observe the nasal mucosa, the inferior nasal concha, and in some cases, the nasal concha. You can see the nasal septum, polyps, and intranasal malformations. In addition, even when there are no structural abnormalities in the nasal cavity, the wider nasal cavity can be intuitively identified. This information is expected to assist in the selection of nostrils. It has not yet been studied whether anesthesiologists select nasal cavity for nasotracheal intubation using prosthesis can affect the occurrence of epistaxis.

The purpose of this study is to determine whether the selection of a nostril for nasotracheal intubation by rhinoscope affects the incidence and severity of epistaxis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II undergoing surgery under nasotracheal intubation

Exclusion Criteria:

* expected difficult intubation based on history, physical examination, weight.
* bleeding tendency
* past history of nasal surgery
* symptom of difficulty of nasal respiration

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
incidence of epistaxis | immediate after intubation
  percentage of the development of epistaxis after nasotracheal intubation
incidence of epistaxis | 5 min after intubation
  percentage of the development of epistaxis after nasotracheal intubation

SECONDARY OUTCOMES:
severity of epistaxis4. severe: interfere intubation by blood | immediate after intubation
  score based on severity of epistaxis will be recorded.
  1: no epistaxis, 2: mild; blood on tube 3. moderate: blood pooling on pharynx
severity of epistaxis | 5 min after intubation
  score based on severity of epistaxis will be recorded.
  1: no epistaxis, 2: mild; blood on tube 3. moderate: blood pooling on pharynx

CONTACTS AND LOCATIONS:
Overall Officials: yun jeong chae, PhD MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou universitiy school of medicine, Suwon, Gyeong-gi Do, South Korea

IPD SHARING:
Plan to Share IPD: No
We will share data when reasonable personal request exist.